CLINICAL TRIAL: NCT03990844
Title: Glycemic Index Evaluation of Noodles Using Functional Ingredients Derived from Food Sources
Brief Title: Glycemic Evaluation of Okra Seed Noodles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Health System (Unknown)
Responsible Party: Principal Investigator, Mei Hui Liu, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/00964
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glucose; Insulin; Ghrelin; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This study is a within-subject cross-over trial to assess the glycemic and insulinemic responses of 0%, 10% and 20% okra-seed enriched noodles in healthy human subjects.
Who Masked: Participant
Masking Description: The investigators will randomized the subjects to consume the noodles at different enrichment levels. Subjects will not know the level of enrichment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0% Okra seed noodle (Placebo Comparator): In this arm, subjects will consume noodles made with 0% okra seed. This serves as a control arm for the study.
  Interventions: Dietary Supplement: Okra seed
- 10% Okra seed noodle (Experimental): In this arm, subjects will consume noodles made with 10% okra seed.
  Interventions: Dietary Supplement: Okra seed
- 20% Okra seed noodle (Experimental): In this arm, subjects will consume noodles made with 10% okra seed.
  Interventions: Dietary Supplement: Okra seed

INTERVENTIONS:
Dietary Supplement: Okra seed — Noodle enriched with 10% and 20% Okra seed flour.

SUMMARY:
In Singapore, the Ministry of Health has declared a "War on Diabetes" and major efforts will be made to develop and deploy programs to prevent diabetes. One of the cornerstones of diabetes management involves dietary modifications to reduce postprandial hyperglycaemia. However, implementation of a low GI diet is highly complex requiring the individual to choose foods from a long list which are primarily based on western consumption patterns. Many foods in the Asian diet, which largely consist of carbohydrates such as white rice, noodles and other flour-based products, are not represented. An alternative solution will require innovative ways to alter commonly available food products that will not only help reduce postprandial glycaemia but also preserve the sensory characteristics of the foods to create a new generation of food products both functional and palatable.

DETAILED DESCRIPTION:
Research has confirmed that a food's glycemic effect cannot be accurately predicted from the type and amount of carbohydrates it contains, as the rate at which the carbohydrates is digested and released into the bloodstream is influenced by many factors such as the food's physical form, its fat, protein and fibre content, and the chemical structure of its carbohydrates. For these reasons, it is possible to produce food from the same group with different effects on blood glucose. Consumption of low glycemic index (GI) food has shown to improve glycemic control, lipid profile and reduce systemic inflammation. However, there are few dietary intervention studies attempting to change the GI of food by changing the staple carbohydrates. In this study, the glycemic index of noodle fortified with Okra seed extract will be determined as compared to a control without the fortification. The fortified noodles have been previously tested to produce lower glycaemic response than noodle without fortification. With noodles being one of the staples to many Singaporeans, noodles fortified with functional ingredients derived from food sources offer a lower GI alternative to the conventional noodles without affecting the people dietary preference.

In the investigator's preliminary study, okra exhibits potential as an anti-diabetic food ingredient in the formulation of low GI staple foods. Indian okra was the most effective overall starch hydrolase inhibitor, inhibiting α-amylase with 50 percent inhibitory concentration (IC50) 2.94 + 0.70 μg/mL and α-glucosidase with IC50 of 23.98 + 1.88 μg/mL. Incorporation of okra seeds into tapioca starch, and rice flour noodles successfully lowered digestibility. To verify in vitro results, human clinical trials is proposed to investigate whether okra seed fortification in noodles successfully retards postprandial hyperglycaemia in humans when consumed.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Chinese male/female age between 21-65 years old
* Healthy as determined by medical history, physical examination and laboratory results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Males and females with stable medical problems that, in the investigator's opinion, will not significantly alter the performance of the biomarker panel, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data.
* Not on any regular medications (western / traditional medicine). Nutritional supplements with established chemical composition that can be ascertained and clearly recorded is acceptable.

However, subjects using traditional medicine (with compositions that cannot be ascertained) will be excluded in this study.

* Have venous access sufficient to allow for blood sampling as per the protocol
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Body mass index of 18 to 25 kg/m2 (male) or 18 to 23 kg/m2 (female).

Exclusion Criteria:

* History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, malignancy or neurological disorders capable of significantly altering the performance of the biomarker panel; or of interfering with the interpretation of data
* Known or ongoing psychiatric disorders within 3 years
* Regularly use known drugs of abuse within 3 years
* Women who are pregnant or lactating
* Have donated blood of more than 500 mL within 4 weeks of study enrolment
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females):

  * 1 unit = 12 oz or 360 mL of beer;
  * 5 oz or 150 mL of wine;
  * 1.5 oz or 45 mL of distilled spirits
* Uncontrolled hypertension (blood pressure >160/100mmHg)
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
* Treatment with any investigational drug, or biological agent within one (1) month of screening or plans to enter into an investigational drug/ biological agent study during the duration of this study
* Known allergy to insulin
* History of bleeding diathesis or coagulopathy
* Any of the following laboratory values at screening:

Fasting glucose >=126mg/dL(>=7mmol/L) or 2 hour post-prandial glucose >=200mg/dL (>=11.1mmol/L)

* Clinically significant (as determined by investigator) abnormalities on laboratory examination that will increase risk to the patient or interfere with data integrity
* Have any other conditions, which, in the opinion of the Investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study
* Significant change in weight (+/- 5%) during the past month
* Known allergy to test food or ingredients used in preparation of test food.
* Subjects with electrical implants/devices such as pacemaker.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in glucose response | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 15 min, 30 min, 45 min, 60 min , 90 min and 120 min.The change in glucose response will be measured by comparing incremental area under the curve (iAUC) after ingestion of noodles.
Change in insulin response | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for glucose analysis at 0 min, 15 min, 30 min, 45 min, 60 min , 90 min and 120 min.The change in insulin response will be measured by comparing incremental area under the curve (iAUC) after ingestion of noodles.

SECONDARY OUTCOMES:
Change in ghrelin level | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for ghrelin analysis at 0 min, 30 min, 60 min , 90 min and 120 min.The change in ghrelin level will be measured by comparing AUC after ingestion of noodles.
Change in glucagon-like peptide 1 (GLP-1) level | 2 hour
  A mixed meal tolerance test will be done to collect blood samples for GLP-1 analysis at 0 min, 30 min, 60 min , 90 min and 120 min.The change in GLP-1 level will be measured by comparing AUC after ingestion of noodles.
Change in satiety rating | 2 hour
  A visual analogue scale (VAS) will be presented to the participants at 0, min, 30 min, 60 min , 90 min and 120 min, to indicate how they feel in response to 4 given statements by marking an "X" on a 100-mm line.
  At time T=15 min, palatability of the treatment was assessed by five characteristics, from bad (0 mm) to good (100 mm). These characteristics were visual appeal, smell, taste, texture, and overall pleasantness of the meal given. Scores were determined by measuring the distance (in mm) from the let starting point of the line to the intersection of the "X". Subjects did not discuss their ratings.The primary outcome was area under the curve (AUC) for responses on the VAS calculated using the trapezoidal rule.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided on a later date.